CLINICAL TRIAL: NCT02484079
Title: Comparative Effectiveness of Hot Versus Cold Snare Polypectomy of Small Colorectal Polyps. A Randomized Controlled Trial
Brief Title: Comparative Effectiveness of Hot Versus Cold Snare Polypectomy of Small Colorectal Polyps
Acronym: HOT/COLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SorlandetHF
Record Dates: First submitted 2015-04-24; First posted 2015-06-29 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2021-12

CONDITIONS: Colonic Polyps; Colorectal Neoplasms; Adenoma
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold polypectomy (Active Comparator): Patients in this arm will have their polyps removed by cold polypectomy, i.e. a metal sling that is closed around the basis of the polyp, and the polyp is cut off.
  After removal there will be taken biopsies from the resection margins, and both the polyp and the biopsies will be examined by a histopathologist to see if the polyp is removed completely.
  Interventions: Procedure: Polypectomy
- Hot polypectomy (Active Comparator): Patients in this arm will have their polyps removed by hot polypectomy, i.e. a metal sling taht is closed around the basis of the polyp, electrical currents is applied, and the polyp is cut off.
  After removal there will be taken biopsies from the resection margins, and both the polyp and the biopsies will be examined by a histopathologist to see if the polyp is removed completely.
  Interventions: Procedure: Polypectomy

INTERVENTIONS:
Procedure: Polypectomy

SUMMARY:
This study aims to investigate the comparative effectiveness between polyp removal with or without electrical current. The investigators want to include 600 polyps in the trial.

It is known that polyps have the potential to develop to cancer if left in situ, but the investigators do not know the best way to remove them completely.

DETAILED DESCRIPTION:
In this study the investigators want to compare to widely used methods for polyp removal; hot and cold snare polypectomy. There has not been performed any big studies on this subject earlier, but current knowledge indicates that hot polypectomy (i.e. with use of electrical current) is somewhat better with regard to complete resection of polyps compared to cold polypectomy (without electrical current).

In this project the patients will be randomized to either hot or cold polypectomy. The investigators will distribute videos of how the polypectomies should be performed, and a gastroenterologist in the project group will instruct the doctors examining the patients to make sure that everyone performs polypectomy according to current guidelines.

The study is designed as a non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient colonoscopy
* Signed, written informed consent
* At least one flat/sessile polyp sized 4-9 mm identified during colonoscopy

Exclusion Criteria:

* Implanted cardiac electro converter
* Severe comorbidity (NYHA 3-4)
* Known coagulopathy (INR > 1,8) or resent use of any of the new oral anti-coagulant medications
* Platelet count < 100
* Resent use of clopidogrel or other non-acetylsalicylic acid platelet inhibitor (Last dose < 5 days before the procedure)
* Previous biopsy or attempt of polypectomy of the polyp considered for inclusion in the trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | Hopefully within 4 weeks, when the histopathologist has examined the biopsies
  We want to measure the rate of polyps that are resected completely, both with biopsies from the margin and the histopathologists evaluation of the resection margins of the polyp itself.

SECONDARY OUTCOMES:
Complications | 4 weeks
  We want to register early (during the procedure) and late (within 4 weeks after the procedure) complications.
  Complications we will record is bleeding/blood in the stool, perforation and patient contact with health care provider
Factors explaining the primary outcome | During the hospital stay and up to 4 weeks.
  Patient characteristics
Factors explaining the primary outcome | During the hospital stay and up to 4 weeks
  Doctor characteristics
Factors explaining the primary outcome | During the hospital stay and up to 4 weeks
  Procedure characteristics
Factors explaining the primary outcome | During the hospital stay and up to 4 weeks
  Histology of polyps, correlation between resection margins and biopsies, correlation between optical and histopathological diagnosis

REFERENCES:
- [Derived] Pedersen IB, Rawa-Golebiewska A, Calderwood AH, Brix LD, Grode LB, Botteri E, Bugajski M, Kaminski MF, Januszewicz W, Odegaard H, Kleist B, Kalager M, Loberg M, Bretthauer M, Hoff G, Medhus A, Holme O. Complete polyp resection with cold snare versus hot snare polypectomy for polyps of 4-9 mm: a randomized controlled trial. Endoscopy. 2022 Oct;54(10):961-969. doi: 10.1055/a-1734-7952. Epub 2022 Jan 10. PMID 35008112